CLINICAL TRIAL: NCT03345758
Title: Department of Critical Care Medicine, Nanjing Zhong-Da Hospital, Southeast University School of Medicine,China;
Brief Title: Long Term Outcome of Extracorporeal Membrane Oxygenation Patients in China
Acronym: ECMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Director, Southeast University, China
Other Study IDs: 20170717
Record Dates: First submitted 2017-10-15; First posted 2017-11-17 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Long-term Outcome; Extracorporeal Membrane Oxygenation
Keywords: respiratory failure, circulatory failure
MeSH Terms: conditions — Respiratory Insufficiency; Shock

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ECMO mode,outcome: ECMO mode includes VV-ECMO and VA-ECMO, outcome includes survive condition , physical and mental health, cognitive function and social adaptation
  Interventions: Other: outcome

INTERVENTIONS:
Other: outcome — telephone to patients to finish SF-36 (the MOS item short from health survey,SF-36)，EQ-5D(EuroQol-5 Dimensions,EQ-5D)， AMT-4（Abbreviated Mental Test-4,AMT-4）and MMSE（Mini-mental State Examination,MMSE） to make assessments of their physical and mental health, cognitive function and social adaptation after discharge

SUMMARY:
Outcomes and Long-term Quality-of-life of Patients requiring Extracorporeal Membrane Oxygenation are not known in china. A prospective study survey will be performed to assess the long-term outcome of these patients.

DETAILED DESCRIPTION:
Patients admitted to ICUs and treated with extracorporeal membrane oxygenation from March 1,2015 to March 1,2019 were screened . Pre-Ecmo clinical parameters(diagnose,APACHE-II, SOFA,indications,expected mortality) and related treatment conditions(duration of ICU stay, duration of ECMO,duration of mechanical ventilation,ventilation conditions,prone ventilation,ECMO complications )will be used to assess the severity and curative effect of these patients.Short Form-36 Health Status Questionnaire,EuroQol-5 Dimensions and St. George's Respiratory Questionnaire(SGRQ) will deliver in these survivors ,which are used to assess the physical and mental health ,as well as the social adaptation. Finally a comprehensive assessment will be obtained to describe the outcomes and long-term quality-of-life of patients treated With ECMO.

ELIGIBILITY:
Inclusion Criteria:

* require extracorporeal membrane oxygenation

Exclusion Criteria:

* irreversible disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated with extracorporeal membrane oxygenation during March,1,2017 to March,1,2019
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
survival rate | August,1,2017-March,1,2020
  survival rate at discharge

SECONDARY OUTCOMES:
Quality of live | August,1,2017-March,1,2020
  Questionnaire：mobility，personal care (washing/dressing)，usual activities，Pain/discomfort，Anxiety/depression
Cognitive function | August,1,2017-March,1,2020
  MMSE Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Qiu, MD, Study Director — professor
Locations (1):
- Nanjing Zhong-Da Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No